CLINICAL TRIAL: NCT00161343
Title: Randomized Controlled Trial of an Group Intervention to Maintain HIV Prevention Gains in Female Adolescents
Brief Title: Maintaining HIV Prevention Gains in Female Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Dianne Morrison-Beedy, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01NR008194 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2009-04

CONDITIONS: HIV Infection; Sexually Transmitted Diseases
Keywords: HIV; Prevention Intervention; Female; Adolescents; STD; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Small interactive groups on preventing HIV infections using an Information-Behavioral Skills-Motivational model
  Interventions: Behavioral: Health Improvement Project for Teens on HIV Prevention
- 2 (Placebo Comparator): Small interactive groups on general health-promotion topics using an Information-Behavioral Skills-Motivational model
  Interventions: Behavioral: Health Improvement Project for Teens on HIV Prevention

INTERVENTIONS:
Behavioral: Health Improvement Project for Teens on HIV Prevention — Comparison of 2 facilitator-led intervention groups: (1) HIV prevention, and (2) general health promotion. Outcome measures: sexual risk behaviors in adolescent girls
  Other Names: HIP Teens

SUMMARY:
In this study, an intervention is tested that is designed to reduced risky sexual behaviors in adolescent females. Study design:

* randomized, controlled study
* participants: 640 girls aged 15-19 years old
* length of follow-up: 1 year after the intervention is completed

Study hypothesis: The experimental condition will significantly reduce risky sexual behaviors in adolescent females as measured by:

* lower incidence of STI's at 6 and 12 months, as compared to baseline
* decreased incidence of risky sexual behaviors
* increased knowledge of the level of risk of certain behaviors
* increased knowledge of safer sexual behaviors that can prevention HIV infection
* increased motivation to reduce sexual risk
* increased behavioral skills to reduce risk of HIV infection

DETAILED DESCRIPTION:
Adolescence is the only age category where the number of females infected with HIV outnumber the number of males. Despite these data, only three randomized controlled trials have evaluated the efficacy of a gender-specific HIV-risk reduction program for adolescent females. The proposed research aims to address this gap in HIV prevention science, and will evaluate the short and longer-term efficacy of a HIV-prevention intervention for adolescent girls. We will recruit 640 adolescent females aged 15 to 19 years from family planning clinics and randomly assign them to one of two conditions: (a) an HIV-risk reduction intervention based on the Information-Motivation-Behavioral Skills (IMB) model (Fisher & Fisher, 1992) or (b) a structurally equivalent health promotion control group (CTL) both supplemented by booster sessions at 3 and 6 months. At a short-term (3-month) follow-up, we hypothesize that IMB participants will increase HIV-related knowledge, motivation, and behavioral skills, and decrease the frequency of risky sexual practices relative to CTL participants. We will reassess all participants at 6 and 12 months to evaluate the longer-term efficacy of the interventions. At these longer-term follow-ups, we hypothesize that IMB participants will demonstrate higher levels of HIV knowledge, motivation, and behavioral skills; decreased risky sexual practices; and decreased rates of STDs (Chlamydia, gonorrhea) relative to the CTL participants. The final aim of the proposed research is to determine whether the constructs in the Information-Motivation-Behavioral Skills (IMB) Model (Fisher & Fisher, 1992), can account for variability in HIV-related behavior. We hypothesize that preventive behavior at 6 and 12 months will be a function of a participant's HIV-related information, motivation, and behavioral skills at the 3-month follow-up, and that information and motivation will be partially mediated by behavioral skills to influence the initiation and maintenance of HIV preventive behavior. The long-term intent of the proposed research is to develop a risk reduction program that can be used by community-based health organizations to reduce the risk of HIV infection among adolescent females.

ELIGIBILITY:
Inclusion Criteria:

* 15-19 years old
* Sexually active in the past 3 months
* Available for follow-up contacts over the next 13 months
* English speaking

Exclusion Criteria:

* Pregnant, or had a baby in the last 3 months
* Married or living with a partner

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 640 (Actual)
Dates: Start 2004-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
rates of STIs | Baseline, 6 and 12 months
computer-assisted survey results | baseline, 1 week, 3, 6, & 12 months
- score on self-report of frequency of risky sexual and substance use behaviors | baseline, 1 week, 3, 6, & 12 months

SECONDARY OUTCOMES:
- score on assessments of information, motivation, and behavioral skills to reduce risk for HIV | baseline, 3, 6, & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dianne C. Morrison-Beedy, Ph.D., RN, Principal Investigator — University of Rochester School of Nursing
Locations (1):
- University of Rochester School of Nursing, Rochester, New York, United States

REFERENCES:
- [Background] Morrison-Beedy D, Aronowitz T, Dyne J, Mkandawire L, Murphy C, Martin J. The nurse clinician as research participant recruiter: experience from a longitudinal intervention study. J N Y State Nurses Assoc. 2001 Fall-Winter;32(2):9-13. PMID 16052902
- [Background] Morrison-Beedy D, Carey MP, Kowalski J, Tu X. Group-based HIV risk reduction intervention for adolescent girls: evidence of feasibility and efficacy. Res Nurs Health. 2005 Feb;28(1):3-15. doi: 10.1002/nur.20056. PMID 15625713
- [Background] Morrison-Beedy D, Carey MP, Aronowitz T. Psychosocial correlates of HIV risk behavior in adolescent girls. J Obstet Gynecol Neonatal Nurs. 2003 Jan-Feb;32(1):94-101. doi: 10.1177/0884217502239806. PMID 12570188
- [Background] Morrison-Beedy D, Carey MP, Aronowitz T, Mkandawire L, Dyne J. An HIV risk-reduction intervention in an adolescent correctional facility: lessons learned. Appl Nurs Res. 2002 May;15(2):97-101. doi: 10.1053/apnr.2002.29530. PMID 11994826
- [Background] Morrison-Beedy D, Carey MP, Aronowitz T, Mkandawire L, Dyne J. Adolescents' input on the development of an HIV risk reduction intervention. J Assoc Nurses AIDS Care. 2002 Jan-Feb;13(1):21-7. doi: 10.1016/S1055-3290(06)60238-0. PMID 11828857
- [Derived] Morrison-Beedy D, Crean HF, Passmore D, Carey MP. Risk reduction strategies used by urban adolescent girls in an HIV prevention trial. Curr HIV Res. 2013 Oct;11(7):559-69. doi: 10.2174/1570162x12666140129110129. PMID 24476350
- [Derived] Morrison-Beedy D, Jones SH, Xia Y, Tu X, Crean HF, Carey MP. Reducing sexual risk behavior in adolescent girls: results from a randomized controlled trial. J Adolesc Health. 2013 Mar;52(3):314-21. doi: 10.1016/j.jadohealth.2012.07.005. Epub 2012 Aug 28. PMID 23299011